CLINICAL TRIAL: NCT01756547
Title: Study to Assess the Efficacy and Safety of Oral Potassium Citrate on the Prevention of Nephrocalcinosis in Extreme Premature.
Acronym: PRENECAL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Juan A. Arnaiz (Other)
Responsible Party: Sponsor-Investigator, Juan A. Arnaiz, Project manager Clinical Trials Unit, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRENECAL
Record Dates: First submitted 2012-12-20; First posted 2012-12-27 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Nephrocalcinosis
Keywords: Nephrocalcinosis; Extreme premature
MeSH Terms: conditions — Nephrocalcinosis | interventions — Potassium Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Potassium citrate (Experimental): Potassium citrate, oral solution contains Tripotassium citrate monohydrate 20 grams, Citric acid monohydrate 4 grams, distilled water 40 ml, and simple syrup 100ml. The solution contained in a bottle of glass that contains 20 ml of 2 meq/ml of potassium and 2.5 meq/ml of citrate. The dose is 0,3ml/kg/day of the solution until the 38-40 weeks of corrected gestational age.
  Interventions: Drug: Potassium Citrate
- Placebo (Placebo Comparator): Oral solution 30ml, that contains distilled water and simple syrup, in the same dose like the active treatment 0,3ml/kg/day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Potassium Citrate — Potassium citrate, oral solution contains Tripotassium citrate monohydrate 20 grams, Citric acid monohydrate 4 grams, distilled water 40 ml, and simple syrup 100ml. The solution contained in a bottle of glass that contains 20 ml of 2 meq/ml of potassium and 2.5 meq/ml of citrate. The dose is 0,3ml/kg/day of the solution until the 38-40 weeks of corrected gestational age or unacceptable toxicity develops.
  Arms: Potassium citrate
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to assess the efficacy and safety of oral potassium citrate on the Prevention of nephrocalcinosis in extreme premature: a clinical trial, randomized, double-blind placebo controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Premature infants of both sexes born at the Hospital Clinic of Barcelona.
2. Corrected gestational age below 32 weeks and lower birth weight 1500gr.
3. Survivors at 7 days old.
4. Clinically stable, in the opinion of the investigator, at the time of inclusion.
5. That, properly informed, parents and / or legal guardians give written consent to allow the participation of the infant in the study and submit to the tests and examinations that it entails

Exclusion Criteria:

1. Renal malformations, cardiac or gastrointestinal prenatal or postnatal diagnosis.
2. Chronic renal failure (serum creatinine> 1.5 mg / dL or an increase of 0.3 mg / dL / day and / or oliguria defined as diuresis <0.5 mL / kg / hour after the first day of life)
3. Treatment with furosemide or dexamethasone
4. Addison's disease.
5. Persistent severe metabolic alkalosis.
6. Impossibility of oral feeding.

Ages: 7 Days to 16 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-12 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
incidence of nephrocalcinosis in extremely preterm infants | 38-40 weeks of corrected gestational age
  incidence of nephrocalcinosis in extremely preterm infants

SECONDARY OUTCOMES:
Determine whether the administration of potassium citrate in extreme premature decreases neonates the levels of calcium and calcium / creatinine ratio in urine in each of the branches of treatment at 38-40 weeks | 38-40 weeks of corrected gestational age
  Determine whether the administration of potassium citrate in extreme premature decreases neonates the levels of calcium and calcium / creatinine ratio in urine in each of the branches of treatment at 38-40 weeks
To determine whether administration of potassium citrate improves the levels of urinary phosphorus, potassium, sodium, citrate, creatinine, oxalate, ratio citrate / calcium , and ph value | 38-40 weeks of corrected gestational age
  To determine whether administration of potassium citrate in extreme premature infants improves the levels of phosphorus, potassium, sodium, citrate, creatinine, oxalate, and ratio citrate / calcium and ph in urine in each treatment arm at the 38-40 weeks.
Determine whether the administration of potassium citrate improves the plasma levels of sodium, potassium, creatinine, calcium, and ph value. | 38-40 weeks of corrected gestational age
  Determine whether the administration of potassium citrate in extreme premature neonates improves the plasma levels of sodium, potassium, creatinine, calcium, and blood ph value in each of the branches of treatment at 38-40 weeks.
To determine the incidence of adverse events and serious adverse events related to study treatment. | 38-40 weeks of corrected gestational age
  To determine the incidence of adverse events and serious adverse events related to study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Botet Mussons, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Barcelona, Spain